CLINICAL TRIAL: NCT03123887
Title: A Retrospective Study to Evaluate the Hematological Remission Rates and Survival Among Chinese Adult Patients With Relapsed or Refractory B-precursor Acute Lymphoblastic Leukemia(ALL)
Brief Title: Evaluate the Hematological Remission Rates and Survival Among Chinese Adult Patients With B-precursor ALL
Acronym: BLING
Status: Completed | Type: Observational
Sponsor: Harbin Hematology and Oncology Institute (Other)
Responsible Party: Principal Investigator, Jun Ma, Chief physician of department of Hematology and Oncology, Harbin Hematology and Oncology Institute
Other Study IDs: TA-ALL-150182
Record Dates: First submitted 2017-04-13; First posted 2017-04-21 (Actual); Last update posted 2017-04-21 (Actual); Status verified 2017-04

CONDITIONS: B-precursor Acute Lymphoblastic Leukemia
MeSH Terms: interventions — Salvage Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- R/r B-precursor ALL: This study selected patients with Relapsed or Refractory (R/r) B-precursor Acute Lymphoblastic Leukemia
  Interventions: Other: salvage therapy

INTERVENTIONS:
Other: salvage therapy — VDC(L)P regimen or High-dose cytarabine based regimen or High-dose methotrexate based regimen or Hyper-CVAD regimen or FLAG (Flu, Ara-C, G-CSF) ± anthracyclines based regimen or Repeated original induction regimen or VDP or other
  Other Names: Ph-PAS

SUMMARY:
Although the response rate by first-line treatment has been improved, most adult patients with relapsed or refractory ALL will eventually relapse with poor outcomes regardless of treatments. To further understand current status of the treatment of adult patients with relapsed or refractory ALL in China, the study retrospectively collected diagnosis and treatment data from ALL patients in 14 centers in China. Primary objective: to estimate the proportion of patients in overall response rate (ORR) for early relapsed or primary refractory Philadelphia chromosome negative (Ph-) B-precursor ALL patients following salvage treatment (i.e., proportion of patients in hematological complete remission [CR] and CR with partial recovery of blood cells [CRh*]); Secondary objectives included: to estimate the proportion of patients in CR, CRh* and CRi(CR/CRh*/CRi) and the duration of CR/CRh*/CRi, overall survival, duration of CR/CRh*and the proportion of patients receiving allogeneic hematopoietic stem cell transplantation (AlloHSCT) for early relapsed/primary refractory Ph-B-precursor ALL patients following salvage treatment; Exploratory objectives included: to estimate the efficacy in late relapsed Ph- B-precursor ALL (first remission duration > 12 months) patients and in Ph+ B-precursor ALL patients and specific subgroup patients following salvage treatment.

DETAILED DESCRIPTION:
Title A Retrospective Study to Evaluate the Hematological Remission Rates and Survival Among Chinese Adult Patients with Relapsed or Refractory B-precursor Acute Lymphoblastic Leukemia (BLING)

Key Words Relapsed or refractory acute lymphoblastic leukemia, complete remission, duration of remission, overall survival, hematopoietic stem cell transplantation

Study Background and Rationale Although the response rate by first-line treatment has been improved, most adult patients with relapsed or refractory ALL will eventually relapse with poor outcome regardless of treatments. In order to improve the diagnosis and treatment level of adult ALL in China, Chinese Society of Hematology and Committee of Hematologic Malignancies of the Chinese Anti-Cancer Association released Expert Consensus on Diagnosis and Treatment of Acute Lymphoblastic Leukemia in Chinese Adult Patients in 2012. However, there is no nationwide multi-center retrospective observational study to evaluate the treatment status of adult patients with R/r ALL (including treatment regimens, and remission rate, overall survival and rate of allogeneic hematopoietic stem cell transplantation of R/r ALL patients following standard salvage chemotherapy), and these data will provide an important reference for further standardization of the treatment of ALL in China, improvement of the prognosis and the research and development of new drugs.

Study questions and Objectives

Primary objectives:

To estimate the proportion of patients in overall response rate (ORR) for early relapsed (a first remission duration of ≤12 months) or primary refractory R/r Philadelphia chromosome negative (Ph-) B-precursor ALL patients following salvage treatment (i.e., proportion of patients in hematological complete remission [CR] and CR with partial recovery of blood cells [CRh*]).

Secondary objectives:

To estimate the proportion of patients in CR, CRh* or CRi for early relapsed/primary refractory Ph-B-precursor ALL patients following salvage treatment (CR/CRh*/CRi) To estimate overall survival (OS) for early relapsed/primary refractory Ph-B-precursor ALL patients following salvage treatment To estimate the duration of CR/CRh* for early relapsed/primary refractory Ph-B-precursor ALL patients following salvage treatment To estimate the duration of CR/CRh*/CRi for early relapsed/primary refractory Ph- B-precursor ALL patients following salvage treatment To estimate the proportion of patients receiving allogeneic hematopoietic stem cell transplantation (AlloHSCT) among early relapsed/primary refractory Ph- B-precursor ALL patients following salvage treatment To examine the potential prognostic factors of early relapsed/primary refractory Ph-B-precursor ALL patients by performing subgroup and regression analyses To estimate overall response rate (CR/CRh*), CR/CRh*/CRi, overall survival (OS), duration of CR/CRh*/CRi, duration of CR/CRh* and the proportion of patients receiving allogeneic hematopoietic stem cell transplantation (AlloHSCT) after CR or CRh* among Ph- B-precursor ALL patients with duration of first CR ≤ 12 months following first salvage treatment

Exploratory objectives:

To estimate the proportion of patients in CR/CRh*, duration of CR/CRh*, proportion of patients in CR/CRh*/CRi, duration of CR/CRh*/CRi, OS and proportion of patients receiving AlloHSCT following salvage treatment for late relapsed (a first remission duration of >12 months) Ph- B-precursor ALL To estimate the proportion of patients in CR/CRh*, duration of CR/CRh*, proportion of patients in CR/CRh*/CRi, duration of CR/CRh*/CRi, OS and the proportion of patients receiving AlloHSCT for Ph+ B-precursor ALL patients and specific subgroup of patients following treatment for R/r B-precursor ALL To examine the potential prognostic factors of late relapsed Ph- B-precursor ALL patients and Ph+ B-precursor ALL patients To describe the types of chemotherapy regimens received and the corresponding efficacy results of main regimens, among patients following primary and salvage treatment for R/r B-precursor ALL Study Design This study was a retrospective study in which data were retrospectively collected from patients with R/r B-precursor ALL in 14 main hematologic malignancy centers in China. Patient subgroups were defined by factors that might influence ORR and OS to better understand their effects on study endpoints.

Subjects and Study Size

The study selected patients with R/r B-precursor ALL meeting inclusion criteria. Specific inclusion criteria were as follows:

Chinese adult patients with R/r B-precursor ALL who had received salvage treatment At least one complete response evaluation results available for salvage treatment With definite Ph chromosome status Age ≥15 years at time of de novo (initial) diagnosis of ALL. For relapsed patients who met the above conditions must also have

1. Evaluable duration of CR by initial therapy, 2. No central nervous system involved at relapsed, 3. No isolated extramedullary relapse.

Patients were divided into 3 analysis sets based on molecular genetic factor and type, and time from initial response to relapse. Ph- Primary Analysis Set included patients who are diagnosed with Ph- disease and meet one of the following criteria: in first relapse or salvage treatment after a first complete remission duration of ≤12 months, or refractory to initial treatment, or relapsed/refractory after first or subsequent salvage treatment, or Relapsed/refractory within 12 months after allogeneic hematopoietic stem cell transplantation (AlloHSCT). The Ph- Late Relapse Analysis Set included patients who had a first remission duration of >12 months and were in first relapse or salvage treatment. The Ph+ Analysis Set included patients who were diagnosed with Ph+ disease.

ELIGIBILITY:
Inclusion Criteria:

* Chinese adult patients with R/r B-precursor ALL who had received salvage treatment
* At least one complete response evaluation results available for salvage treatment
* With definite Ph chromosome status
* Age ≥15 years at time of de novo (initial) diagnosis of ALL.
* For relapsed patients who met the above conditions must also have
* Evaluable duration of CR by initial therapy
* No central nervous system involved at relapsed
* No isolated extramedullary relapse Patients were divided into 3 analysis sets based on molecular genetic factor and type, and time from initial response to relapse.
* Ph- Primary Analysis Set included patients who are diagnosed with Ph- disease and meet one of the following criteria:
* in first relapse or salvage treatment after a first complete remission duration of ≤12 months, or refractory to initial treatment, or relapsed/refractory after first or subsequent salvage treatment, or Relapsed/refractory within 12 months after alloHSCT.
* The Ph- Late Relapse Analysis Set included patients who had a first remission duration of >12 months and were in first relapse or salvage treatment.
* The Ph+ Analysis Set included patients who were diagnosed with Ph+ disease.

Exclusion Criteria:

-

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Relapsed or Refractory B-precursor Acute Lymphoblastic Leukemia
Sampling Method: Probability Sample
Enrollment: 632 (Actual)
Dates: Start 2015-07-10 (Actual); Primary Completion 2016-06-03 (Actual); Study Completion 2016-10-10 (Actual)

PRIMARY OUTCOMES:
overall response rate | up to 3 years
  overall response rate after the last salvage therapy, i.e., CR/CRh*. CR is generally defined as no blasts in peripheral blood, absence of extramedullary leukemia, full recovery of peripheral blood counts, ≤ 5% blasts in the bone marrow, ANC > 1.0×109/L, PLT > 100×109/L, no relapse within 4 weeks. CRh* was CR with partial recovery of peripheral blood counts, ANC > 0.5×109/L, PLT > 50×109/L, with other conditions meeting the criteria for CR

SECONDARY OUTCOMES:
proportion of patients in CR, CRh* or CRi | up to 3 years
  the proportion of patients in CR, CRh* or CRi for early relapsed/primary refractory Ph- B-precursor ALL patients following last salvage treatment
overall survival | up to 3 years
  overall survival (OS) for early relapsed/primary refractory Ph- B-precursor ALL patients after CR or CRh* achieved
duration of remission (CR/CRh*, CR/CRh*/CRi) | up to 3 years
  duration of remission (CR/CRh*, CR/CRh*/CRi) for early relapsed/primary refractory Ph- B-precursor ALL patients after CR or CRh* achieved
proportion of patients receiving allogeneic hematopoietic stem cell transplantation | up to 3 years
  the proportion of patients receiving allogeneic hematopoietic stem cell transplantation (AlloHSCT) among early relapsed/primary refractory Ph- B-precursor ALL patients following salvage treatment
overall survival | up to 3 years
  overall survival (OS) among R/r Ph- B-precursor ALL patients after achieving CR or CRh* after the first salvage therapy
duration of CR/CRh*/CRi | up to 3 years
  duration of CR/CRh* among R/r Ph- B-precursor ALL patients after achieving CR or CRh* after the first salvage therapy
the proportion of patients receiving allogeneic hematopoietic stem cell transplantation (AlloHSCT) | up to 3 years
  the proportion of patients receiving allogeneic hematopoietic stem cell transplantation (AlloHSCT) after CR or CRh* achieved among R/r Ph- B-precursor ALL patients after achieving CR or CRh* after the first salvage therapy
Complete Response | up to 3 years
  Complete Response among R/r Ph- B-precursor ALL patients after achieving CR or CRh* after the first salvage therapy
Complete Response with incomplete recovery of blood cells | up to 3 years
  Complete Response with incomplete recovery of blood cells among R/r Ph- B-precursor ALL patients after achieving CR or CRh* after the first salvage therapy
Complete Response with partial recovery of blood cells | up to 3 years
  Complete Response with partial recovery of blood cells among R/r Ph- B-precursor ALL patients after achieving CR or CRh* after the first salvage therapy
duration of CR/CRh* | up to 3 years
  duration of CR/CRh* with partial recovery of blood cells among R/r Ph- B-precursor ALL patients after achieving CR or CRh* after the first salvage therapy

CONTACTS AND LOCATIONS:
Overall Officials: Jun Ma, director, Study Chair — Institute of Harbin Hematology Oncology
Locations (1):
- Institute of Harbin Hematology Oncology, Harbin, Heilongjiang, China

IPD SHARING:
Plan to Share IPD: No
To protect the privacy of individual who participate in this trial we would not share the individual data with other researchers

REFERENCES:
- [Background] Bassan R, Gatta G, Tondini C, Willemze R. Adult acute lymphoblastic leukaemia. Crit Rev Oncol Hematol. 2004 Jun;50(3):223-61. doi: 10.1016/j.critrevonc.2003.11.003. PMID 15182827
- [Background] Fielding AK, Richards SM, Chopra R, Lazarus HM, Litzow MR, Buck G, Durrant IJ, Luger SM, Marks DI, Franklin IM, McMillan AK, Tallman MS, Rowe JM, Goldstone AH; Medical Research Council of the United Kingdom Adult ALL Working Party; Eastern Cooperative Oncology Group. Outcome of 609 adults after relapse of acute lymphoblastic leukemia (ALL); an MRC UKALL12/ECOG 2993 study. Blood. 2007 Feb 1;109(3):944-50. doi: 10.1182/blood-2006-05-018192. Epub 2006 Oct 10. PMID 17032921
- [Background] Gokbuget N, Stanze D, Beck J, Diedrich H, Horst HA, Huttmann A, Kobbe G, Kreuzer KA, Leimer L, Reichle A, Schaich M, Schwartz S, Serve H, Starck M, Stelljes M, Stuhlmann R, Viardot A, Wendelin K, Freund M, Hoelzer D; German Multicenter Study Group for Adult Acute Lymphoblastic Leukemia. Outcome of relapsed adult lymphoblastic leukemia depends on response to salvage chemotherapy, prognostic factors, and performance of stem cell transplantation. Blood. 2012 Sep 6;120(10):2032-41. doi: 10.1182/blood-2011-12-399287. Epub 2012 Apr 4. PMID 22493293
- [Background] Jabbour EJ, Faderl S, Kantarjian HM. Adult acute lymphoblastic leukemia. Mayo Clin Proc. 2005 Nov;80(11):1517-27. doi: 10.4065/80.11.1517. PMID 16295033
- [Background] Larson RA. Acute lymphoblastic leukemia: older patients and newer drugs. Hematology Am Soc Hematol Educ Program. 2005:131-6. doi: 10.1182/asheducation-2005.1.131. PMID 16304370
- [Background] Le QH, Thomas X, Ecochard R, Iwaz J, Lheritier V, Michallet M, Fiere D. Proportion of long-term event-free survivors and lifetime of adult patients not cured after a standard acute lymphoblastic leukemia therapeutic program: adult acute lymphoblastic leukemia-94 trial. Cancer. 2007 May 15;109(10):2058-67. doi: 10.1002/cncr.22632. PMID 17407135
- [Background] Liu L, Jiao W, Zhang Y, Qu Q, Li X, Wu D. Efficacy of low-dose cytarabine and aclarubicin in combination with granulocyte colony-stimulating factor (CAG regimen) compared to Hyper-CVAD regimen as salvage chemotherapy in relapsed/refractory Philadelphia chromosome-negative acute lymphoblastic leukemia. Leuk Res. 2015 Mar;39(3):323-8. doi: 10.1016/j.leukres.2015.01.003. Epub 2015 Jan 16. PMID 25638269
- [Background] Oriol A, Vives S, Hernandez-Rivas JM, Tormo M, Heras I, Rivas C, Bethencourt C, Moscardo F, Bueno J, Grande C, del Potro E, Guardia R, Brunet S, Bergua J, Bernal T, Moreno MJ, Calvo C, Bastida P, Feliu E, Ribera JM; Programa Espanol de Tratamiento en Hematologia Group. Outcome after relapse of acute lymphoblastic leukemia in adult patients included in four consecutive risk-adapted trials by the PETHEMA Study Group. Haematologica. 2010 Apr;95(4):589-96. doi: 10.3324/haematol.2009.014274. Epub 2010 Feb 9. PMID 20145276
- [Background] Pui CH, Evans WE. Acute lymphoblastic leukemia. N Engl J Med. 1998 Aug 27;339(9):605-15. doi: 10.1056/NEJM199808273390907. No abstract available. PMID 9718381
- [Background] Thomas DA, Kantarjian H, Smith TL, Koller C, Cortes J, O'Brien S, Giles FJ, Gajewski J, Pierce S, Keating MJ. Primary refractory and relapsed adult acute lymphoblastic leukemia: characteristics, treatment results, and prognosis with salvage therapy. Cancer. 1999 Oct 1;86(7):1216-30. doi: 10.1002/(sici)1097-0142(19991001)86:73.0.co;2-o. PMID 10506707
- [Background] Yan CH, Wang JZ, Liu DH, Xu LP, Chen H, Liu KY, Huang XJ. Chemotherapy followed by modified donor lymphocyte infusion as a treatment for relapsed acute leukemia after haploidentical hematopoietic stem cell transplantation without in vitro T-cell depletion: superior outcomes compared with chemotherapy alone and an analysis of prognostic factors. Eur J Haematol. 2013 Oct;91(4):304-14. doi: 10.1111/ejh.12168. Epub 2013 Aug 17. PMID 23837640